CLINICAL TRIAL: NCT04468282
Title: Bioequivalence Study of Vigabatrin ORPHELIA Pharma 500mg Soluble Tablets and SabrilTM 500mg Granules for Oral Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orphelia Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ORP-VGB-I-a; 2017-000038-67 (EudraCT Number)
Record Dates: First submitted 2020-03-27; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Therapeutic Equivalency

STUDY DESIGN:
Intervention Model Description: The study was an open label, randomized, crossover, 2 periods study in 20 healthy male/female volunteers. Subjects received 500 mg of the new formulation of soluble tablets vigabatrin or Sabril TM, as single oral administration in 2 different study periods depending on the randomization, with a 7-days wash out period between administrations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VGB-ST (Experimental): Name of the compound: Vigabatrin ORPHELIA Pharma (VGB-ST) Pharmaceutical form: Soluble tablet Dose per administration: 500 mg Timing for administration: Single oral administration on P1D1 or P2D1 according to randomization.
  Batch N°: 16.92.042 (expiry date: 31.05.2017)
  Interventions: Drug: VGB-ST
- Sabril (Active Comparator): Name of the compound: Sabril (vigabatrin) Pharmaceutical form: granules (sachet) Dose per administration: 500 mg Timing for administration: Single oral administration on P1D1 or P2D1 according to randomization.
  Batch N°: 6810 (expiry date: 31.05.2019)
  Interventions: Drug: VGB-ST

INTERVENTIONS:
Drug: VGB-ST — Single oral administration of 500 mg VGB-ST
  Other Names: vigabatrin soluble tablets; Kigabeq

SUMMARY:
Methodology:

The study was an open label, randomized, crossover, 2 periods study in 20 healthy male/female volunteers. Subjects received 500 mg of the new formulation of soluble tablets vigabatrin or Sabril, as single oral administration in 2 different study periods depending on the randomization, with a 7-days wash out period between administrations

DETAILED DESCRIPTION:
Objectives:

Primary objective:

Evaluate bioequivalence between a new paediatric formulation of vigabatrin (VGB-ST) and Sabril granules for oral administration.

Secondary objective:

* Define pharmacokinetic parameters of the new paediatric formulation soluble tablets of vigabatrin (VGB-ST)
* Assess the safety of the new formulation of soluble tablets VGB-ST versus Sabril

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subject, aged between 18 and 50 years inclusive;
2. Females of childbearing potential/Sexually active males with partner of childbearing potential: commitment to consistently and correctly use an acceptable method of birth control (oral, transdermal, systemic or implant contraception birth control, intrauterine devices, diaphragm, condoms or abstinence) for the duration of the trial and for 1 month after the last study drug administration; Females of non-childbearing potential: either surgically sterilized or at least 1 year postmenopausal (amenorrhoea duration at least 12 months);
3. Non breast-feeding female and negative pregnancy test at screening baseline;
4. Non-smoker subject or smoker of not more than 5 cigarettes per day;
5. Body Mass Index (BMI) between 18,5 and 25 kg/m2 inclusive;
6. Considered as healthy after a comprehensive clinical assessment (detailed medical history and complete physical examination);
7. Normal Blood Pressure (BP) and Heart Rate (HR) at the screening visit after 10 minutes in supine position
8. Normal ECG recording on a 12-lead ECG at the screening visit
9. Laboratory parameters within the normal range of the laboratory (hematological, blood chemistry tests, urinalysis). Individual values out of the normal range could be accepted if judged clinically non relevant by the Investigator;
10. Normal dietary habits;
11. Signing a written informed consent prior to selection;
12. Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.

Exclusion Criteria:

1. Any history or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, haematological, neurologic, psychiatric, systemic, infectious disease or psychiatric disorders;
2. Frequent headaches and / or migraine, recurrent nausea and / or vomiting;
3. History of abnormal vision (e.g. reduced visual field, retinopathy, etc…);
4. Abnormal visual field recorded during the inclusion period;
5. Evidence of any clinically significant acute or chronic disease;
6. Symptomatic hypotension whatever the decrease of blood pressure or asymptomatic postural hypotension defined by a decrease in SBP or DBP equal to or greater than 20 mmHg within two minutes when changing from the supine to the standing position;
7. Surgery or blood donation (including in the frame of a clinical trial) within 2 months before administration;
8. General anaesthesia within 3 months before administration;
9. Presence or history of drug hypersensitivity, asthma or allergic disease diagnosed and treated by a physician;
10. Inability to abstain from intensive muscular effort;
11. No possibility of contact in case of emergency;
12. Any drug intake (except paracetamol or contraception) during the last month prior to the first administration;
13. History or presence of drug or alcohol abuse (alcohol consumption > 40 grams / day);
14. Excessive consumption of beverages containing xanthine bases (> 4 cups or glasses / day);
15. Positive Hepatitis B surface (HBs) antigen or anti Hepatitis C Virus (HCV) antibody (not including HSV), or positive results for Human Immunodeficiency Virus (HIV) 1 or 2 tests;
16. Positive results of screening for drugs of abuse;
17. Subject who, in the judgment of the Investigator, was likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development;
18. Exclusion period of a previous study;
19. Administrative or legal supervision;
20. Subject who would receive more than 4500 euros as indemnities for his participation in biomedical research within the 12 last months, including the indemnities for the present study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

PRIMARY OUTCOMES:
Primary pharmacokinetic parameters (Bioequivalence) | day 1 or 2
  The following pharmacokinetic parameters were determined from S(+) enantiomer of vigabatrin plasma concentrations: Cmax
Primary pharmacokinetic parameters (Bioequivalence) | day 1 or 2
  The following pharmacokinetic parameters were determined from S(+) enantiomer of vigabatrin plasma concentrations: AUC0-t

SECONDARY OUTCOMES:
Secondary pharmacokinetic parameters | day 1 or 2
  The following pharmacokinetic parameters were determined from S(+) enantiomer of vigabatrin plasma concentrations: AUC0-inf
Secondary pharmacokinetic parameters | day 1 or 2
  The following pharmacokinetic parameters were determined from S(+) enantiomer of vigabatrin plasma concentrations: tmax
Secondary pharmacokinetic parameters | day 1 or 2
  The following pharmacokinetic parameters were determined from S(+) enantiomer of vigabatrin plasma concentrations: λ
Secondary pharmacokinetic parameters | day 1 or 2
  The following pharmacokinetic parameters were determined from S(+) enantiomer of vigabatrin plasma concentrations: t1/2
Secondary pharmacokinetic parameters | day 1 or 2
  The following pharmacokinetic parameters were determined from S(+) enantiomer of vigabatrin plasma concentrations: residual area

CONTACTS AND LOCATIONS:
Overall Officials: PharmD PharmD, PhD, Study Director — Orphelia Pharma
Locations (1):
- Eurofins Optimed, Gières, France

IPD SHARING:
Plan to Share IPD: No